CLINICAL TRIAL: NCT03230084
Title: Use of a Home-based Urinary Pregnanediol 3-glucuronide (PDG) Test to Confirm Ovulation
Brief Title: Use of a Home-based PDG Urine Test to Confirm Ovulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Rene Leiva, MD (Unknown); Bruyere Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: M16-17-027
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-07

CONDITIONS: Infertility, Female
Keywords: Infertility; Ovulation; Pregnanediol 3-glucuronide; Progesterone; Urine dipstick test; Feasibility study; Fertile period; Menstrual cycle; Natural family planning; Fertility awareness methods
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Urine PDG test (Experimental): Urine pregnanediol 3-glucuronide (PDG) test strip
  Interventions: Device: Urine PDG test

INTERVENTIONS:
Device: Urine PDG test — Urine dipstick test that detects the presence of the urinary metabolite of progesterone, PDG.

SUMMARY:
Infertility affects many people in Ontario and carries a significant amount of emotional, physical and financial burden to those who experience it. Knowing when a woman ovulates is important for improving a couple's chance to become pregnant naturally and for learning about fertility problems, such as infertility, irregular menses, and hormonal disorders.

Currently, there are two reliable methods to confirm ovulation: a trans-vaginal ultrasound or a blood test for progesterone, which is a hormone that only rises sharply after ovulation. However, both are time consuming and expensive. Recently, an inexpensive, home-based urine test strip has been developed to confirm ovulation. The test strip works by measuring urine for a marker of Progesterone, called pregnanediol-3a-glucuronide (PDG).

The purpose of this feasibility study is to follow the use of this home-based PDG urinary test strip over the course of one menstrual cycle in 25 female participants. The results of the urine test strip will then be compared to a Progesterone blood test. Participants will be recruited from the general Ottawa, Ontario area The ultimate aim of this study is to provide information for the design of a larger study to determine the accuracy of the PDG urinary test strip. If shown to be as effective in confirming ovulation, this test would provide substantial cost saving to the Ontario health care system and a much more convenient way for women and clinicians to confirm ovulation and determine if women are fertile.

DETAILED DESCRIPTION:
Infertility affects many people in Ontario and carries a significant amount of emotional, physical and financial burden to those who experience it. More specifically, it impacts the couple's quality of life and can have detrimental effects related to marital conflicts, couple burnout and psychological disorders including a lack of confidence and depression.

As part of the standard evaluation of infertility, ovulatory function assessment is a fundamental step. Confirmation that ovulation has actually occurred can only be determined by performing a serum Progesterone test or by using the gold standard, serial transvaginal ultrasound. However, both of these investigations require visits to a physician, specialized laboratory testing, and in the case of ultrasound are often prohibitive due to its high costs and logistical demands.

In the female body, levels of Progesterone are low in the first half of the menstrual cycle. After the ovary releases an egg (ovulation) the corpus luteum produces high levels of Progesterone. Pregnanediol-3a-glucuronide (PDG) is the major urine metabolite of Progesterone. An inexpensive, home-based PDG urine test strip to confirm ovulation has recently been developed. The PDG test measures the presence of PDG in urine, which has been shown to directly correlate with the presence Progesterone in serum (blood). According to GLOWM (The Global Library of Women's Medicine) PDG levels in urine typically rise 24-36 hours after ovulation.

Although there also exists a home-based electronic hormone monitor for measuring urinary PDG, it is not widely available and is very time-consuming for women. Newer methods to monitor PDG using a simple urinary test strip that are less time consuming would be a welcome addition to the evaluation of infertility. Additionally, urinary hormonal tests have been proven to be easy and useful adjuncts to natural fertility markers.

The primary purpose of this feasibility study is to evaluate the use of the PDG urine test in a clinical setting to determine its accuracy to confirm ovulation when compared to the serum Progesterone test. This study will follow the use of the PDG urinary test strip over the course of one menstrual cycle in 25 female participants. In order to obtain participants, this study will use a non-probability sample using an initiation to volunteer technique for women in the general Ottawa area. The ultimate aim of this study is to provide information for the design of a larger study to determine the accuracy of the PDG urinary test strip.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 42 years
* Have had a menstrual cycle length of 25-35 days for the past 3 months
* Are able to provide informed consent
* Are willing to complete a trial diary

Exclusion Criteria:

* Have current or recent (in the past 6 months) use of any hormonal contraception (e.g. the Pill, Norplant, Depo Provera injections)
* Have current or recent (in the past 6 months) breastfeeding
* Have use of emergency contraception (e.g. the morning after pill or Plan B) in the past two menstrual cycles
* Cannot medically receive frequent blood tests, for example due to a blood clotting disorder
* Are pregnant at the time of enrollment to study
* Plan to donate blood during the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the PDG urine test strip | 1 month
  The sensitivity will be estimated as the proportion of true positives cycles, that is, cycles with appropriate recognition of the post-ovulatory phase. The specificity will be estimated as the proportion of true negatives cycles, that is, cycles with appropriate recognition of the pre-ovulatory phase.

SECONDARY OUTCOMES:
Frequency of protocol violation | 1 month
  Percentage of participants who violated protocol to show acceptability of study design to participants.
Frequency of positive responses versus negative responses about the study procedures | 1 month
  Ratio of positive responses to negative responses in the feedback questionnaire given to participants concerning the study protocol.
Frequency of positive responses versus negative responses on the study product | 1 month
  Ratio of positive responses to negative responses in the feedback questionnaire given to participants concerning the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Leiva, MD, Principal Investigator — Bruyère Health Research Institute.
Locations (1):
- Bruyere Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ecochard R, Leiva R, Bouchard T, Boehringer H, Direito A, Mariani A, Fehring R. Use of urinary pregnanediol 3-glucuronide to confirm ovulation. Steroids. 2013 Oct;78(10):1035-40. doi: 10.1016/j.steroids.2013.06.006. Epub 2013 Jul 4. PMID 23831784
- [Background] Messerlian C, Fishman JR. Less is more: improving outcomes and cutting costs to Quebec's assisted reproduction program. CMAJ. 2014 Apr 1;186(6):405-6. doi: 10.1503/cmaj.131672. Epub 2014 Mar 3. No abstract available. PMID 24591273
- [Background] Brown JB. Types of ovarian activity in women and their significance: the continuum (a reinterpretation of early findings). Hum Reprod Update. 2011 Mar-Apr;17(2):141-58. doi: 10.1093/humupd/dmq040. Epub 2010 Oct 5. PMID 20923873
- [Background] Vigil P, Ceric F, Cortes ME, Klaus H. Usefulness of monitoring fertility from menarche. J Pediatr Adolesc Gynecol. 2006 Jun;19(3):173-9. doi: 10.1016/j.jpag.2006.02.003. PMID 16731410
- [Background] Bushnik T, Cook JL, Yuzpe AA, Tough S, Collins J. Estimating the prevalence of infertility in Canada. Hum Reprod. 2012 Mar;27(3):738-46. doi: 10.1093/humrep/der465. Epub 2012 Jan 17. PMID 22258658
- [Background] Ghavi F, Jamale S, Mosalanejad L, Mosallanezhad Z. A Study of Couple Burnout in Infertile Couples. Glob J Health Sci. 2015 Aug 6;8(4):158-65. doi: 10.5539/gjhs.v8n4p158. PMID 26573033
- [Background] Evans-Hoeker E, Pritchard DA, Long DL, Herring AH, Stanford JB, Steiner AZ. Cervical mucus monitoring prevalence and associated fecundability in women trying to conceive. Fertil Steril. 2013 Oct;100(4):1033-1038.e1. doi: 10.1016/j.fertnstert.2013.06.002. Epub 2013 Jul 11. PMID 23850303
- [Background] Robinson JE, Wakelin M, Ellis JE. Increased pregnancy rate with use of the Clearblue Easy Fertility Monitor. Fertil Steril. 2007 Feb;87(2):329-34. doi: 10.1016/j.fertnstert.2006.05.054. Epub 2006 Oct 30. PMID 17074329
- [Background] Leiva R, Bouchard T, Boehringer H, Abulla S, Ecochard R. Random serum progesterone threshold to confirm ovulation. Steroids. 2015 Sep;101:125-9. doi: 10.1016/j.steroids.2015.06.013. Epub 2015 Jun 22. PMID 26111590
- [Background] Practice Committee of American Society for Reproductive Medicine. Diagnostic evaluation of the infertile female: a committee opinion. Fertil Steril. 2012 Aug;98(2):302-7. doi: 10.1016/j.fertnstert.2012.05.032. Epub 2012 Jun 13. PMID 22698637
- [Background] Practice Committee of American Society for Reproductive Medicine in collaboration with Society for Reproductive Endocrinology and Infertility. Optimizing natural fertility: a committee opinion. Fertil Steril. 2013 Sep;100(3):631-7. doi: 10.1016/j.fertnstert.2013.07.011. PMID 23993665
- [Background] Stanford JB. Revisiting the fertile window. Fertil Steril. 2015 May;103(5):1152-3. doi: 10.1016/j.fertnstert.2015.02.015. Epub 2015 Mar 13. No abstract available. PMID 25772771
- [Background] Leiva R, Burhan U, Kyrillos E, Fehring R, McLaren R, Dalzell C, Tanguay E. Use of ovulation predictor kits as adjuncts when using fertility awareness methods (FAMs): a pilot study. J Am Board Fam Med. 2014 May-Jun;27(3):427-9. doi: 10.3122/jabfm.2014.03.130255. PMID 24808123
- [Background] Ecochard R, Boehringer H, Rabilloud M, Marret H. Chronological aspects of ultrasonic, hormonal, and other indirect indices of ovulation. BJOG. 2001 Aug;108(8):822-9. doi: 10.1111/j.1471-0528.2001.00194.x. PMID 11510707
- [Background] Ecochard R, Duterque O, Leiva R, Bouchard T, Vigil P. Self-identification of the clinical fertile window and the ovulation period. Fertil Steril. 2015 May;103(5):1319-25.e3. doi: 10.1016/j.fertnstert.2015.01.031. Epub 2015 Feb 24. PMID 25724738
- [Background] Blackwell LF, Vigil P, Alliende ME, Brown S, Festin M, Cooke DG. Monitoring of ovarian activity by measurement of urinary excretion rates using the Ovarian Monitor, Part IV: the relationship of the pregnanediol glucuronide threshold to basal body temperature and cervical mucus as markers for the beginning of the post-ovulatory infertile period. Hum Reprod. 2016 Feb;31(2):445-53. doi: 10.1093/humrep/dev303. Epub 2015 Dec 17. PMID 26677961
- [Background] Sauer MV, Paulson RJ. Utility and predictive value of a rapid measurement of urinary pregnanediol glucuronide by enzyme immunoassay in an infertility practice. Fertil Steril. 1991 Nov;56(5):823-6. doi: 10.1016/s0015-0282(16)54649-4. PMID 1936313
- [Background] Denari JH, Farinati Z, Casas PR, Oliva A. Determination of ovarian function using first morning urine steroid assays. Obstet Gynecol. 1981 Jul;58(1):5-9. PMID 7195531
- [Background] Adlercreutz H, Brown J, Collins W, Goebelsman U, Kellie A, Campbell H, Spieler J, Braissand G. The measurement of urinary steroid glucuronides as indices of the fertile period in women. World Health Organization, Task Force on Methods for the Determination of the Fertile Period, special programme of research, development and research training in human reproduction. J Steroid Biochem. 1982 Dec;17(6):695-702. doi: 10.1016/0022-4731(82)90573-8. PMID 7176659
- [Background] Sauer MV, Paulson RJ, Chenette P, Frederick J, Stanczyk FZ. Effect of hydration on random levels of urinary pregnanediol glucuronide. Gynecol Endocrinol. 1990 Sep;4(3):145-9. doi: 10.3109/09513599009009801. PMID 2284979
- [Background] Stirnemann JJ, Samson A, Bernard JP, Thalabard JC. Day-specific probabilities of conception in fertile cycles resulting in spontaneous pregnancies. Hum Reprod. 2013 Apr;28(4):1110-6. doi: 10.1093/humrep/des449. Epub 2013 Jan 22. PMID 23340057
- [Background] Wesselink AK, Wise LA, Hatch EE, Rothman KJ, Mikkelsen EM, Stanford JB, McKinnon CJ, Mahalingaiah S. Menstrual cycle characteristics and fecundability in a North American preconception cohort. Ann Epidemiol. 2016 Jul;26(7):482-487.e1. doi: 10.1016/j.annepidem.2016.05.006. Epub 2016 May 31. PMID 27449569
- [Background] Bigelow JL, Dunson DB, Stanford JB, Ecochard R, Gnoth C, Colombo B. Mucus observations in the fertile window: a better predictor of conception than timing of intercourse. Hum Reprod. 2004 Apr;19(4):889-92. doi: 10.1093/humrep/deh173. Epub 2004 Feb 27. PMID 14990542
- [Derived] Leiva R, McNamara-Kilian M, Niezgoda H, Ecochard R, Bouchard T. Pilot observational prospective cohort study on the use of a novel home-based urinary pregnanediol 3-glucuronide (PDG) test to confirm ovulation when used as adjunct to fertility awareness methods (FAMs) stage 1. BMJ Open. 2019 May 27;9(5):e028496. doi: 10.1136/bmjopen-2018-028496. PMID 31133596
- See also: : As couples search for satisfactory forms of contraception, some 'rediscover' a traditional method; others are introduced to birth control by an unconventional messenger. — http://articles.latimes.com/1993-01-07/news/vw-935_1_birth-controlmethods
- See also: Fertility problems: assessment and treatment — https://www.nice.org.uk/guidance/cg156